CLINICAL TRIAL: NCT06973746
Title: Effect of the "Sitting Out of Bed in an Arm-chair Position" in ICU on Functional Recovery Among Ventilated Patients: a Prospective Randomized Controlled Trial
Brief Title: Effect of the "Sitting Out of Bed in an Arm-chair Position" in ICU on Functional Recovery Among Ventilated Patients
Acronym: STORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUO-2024-17
Record Dates: First submitted 2025-04-28; First posted 2025-05-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: ICU Acquired Weakness
Keywords: mechanical ventilation; ICU Acquired Weakness; Arm Chair; Sitting; Early mobility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sitting out of bed in an arm-chair position (Experimental)
  Interventions: Other: sitting out of bed in an arm-chair position
- No chair position (No Intervention)

INTERVENTIONS:
Other: sitting out of bed in an arm-chair position — Once the patient has been awake with a RASS score between -1 and +1 for more than 12 hours, he or she must be placed in a chair (by any means) every day for a minimum of 30 minutes until "discharge" from intensive care (or until D28, depending on which comes first), unless there are transient contraindications. If the patient is unable to signal his or her wish to stop the chair session, the criteria for intolerance will be sought and the patient placed in the chair, but in all cases the chair session will not exceed 4 hours.
  Arms: sitting out of bed in an arm-chair position

SUMMARY:
Chair positioning is one of a series of early mobilization techniques. At present, this technique, which involves moving a patient out of the resuscitation bed, can be performed passively or actively. It does not constitute a rehabilitative act as such, but it is considered in common paradigms as a technique to improve "the patient's breathing and strength".

However, recommendations issued in 2013 by the Society of intensive care physiotherapy and the society "Société de réanimation de langue française (SRLF)", reveal that this chair position cannot be recommended with a high grade.

The aim of the investigators is therefore to break down this early mobilization process in intensive care, to find out whether the armchair is an indispensable tool for improving functional and muscular processes.

The research hypothesis is therefore as follows:

"Early armchairing of the resuscitation patient, improves functional recovery compared to a conservative positioning strategy (sitting in bed)."

ELIGIBILITY:
Inclusion Criteria:

1. Patient > 18 years old
2. Patient on invasive mechanical ventilation for more than 24 hours
3. Patient in recovery phase with a RASS score greater than "-3" for more than 12 hours
4. Stay expected to last 48 hours
5. Patient has never been placed in a chair during this hospitalization in intensive care.
6. Fragility score < 6, during the month preceding admission to intensive care
7. Patient (or support person/relative if patient is unable to participate) who has agreed to take part in the study.

Exclusion Criteria:

1. Patient with an absolute and non-resolving contraindication to chair positioning

   1. Fracture or orthopedic disorder contraindicating mobilization out of bed
   2. Obesity with body mass index greater than 45 kg/cm2
   3. Sacral eschar stage greater than 2
2. Patient using a wheelchair for mobility (i.e. paraplegic patient or patient with progressive neurological pathology).
3. Patient treated with veno-venous or veno-arterial ECMO at the time of screening.
4. Moribund patient
5. Encephalic death
6. Acute polyradiculoneuritis (Guillain-Barré syndrome)
7. Myasthenia
8. Patient treated by continuous hemodialysis or hemofiltration for more than 72 hours following the onset of awakening.
9. Complete transmetatarsal or higher amputation of one or both lower limbs.
10. Protected person (under guardianship or curatorship)
11. Person under court protection
12. Person not affiliated to a social security scheme
13. Pregnant or breast-feeding woman
14. Patient already included in the study
15. Patient taking part in an interventional clinical study, the aim of which is to show an improvement in functional level on discharge from the intensive care unit or which focuses on the theme of early rehabilitation in the intensive care unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Functional level on "discharge" from intensive care | On discharge from intensive care or day 28 (depending on which comes first)
  Functional level at "discharge" from the intensive care unit measured by the Physical Function ICU Test scored (PFIT-s).
  Minimum value = 0 , meaning worse functionnal status Maximum value = 12, meaning better functionnal status

SECONDARY OUTCOMES:
ICU Mobility scale | Day 28
  Maximum level of mobility achieved Minimum value = 0, meaning "no mobility" Maximum value = 10, meaning "walking without assistance"
MRC sum score | Day 28
  Presence of muscular weakness acquired in intensive care Minimum value = 0, meaning "no muscular contraction" Maximum value = 60, meaning "normal muscular force"
Length of stay in intensive care unit | Day 28
Ventilator free days | Day 28
  Number of days without invasive mechanical ventilation
Mortality rate | Day 28
Total length of hospital stay | Day 28
Mortality | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FOSSAT, Principal Investigator — CHU Orléans
Locations (11):
- France (11):
  - Centre Hospitalier Universitaire d'Orléans, Orléans, Centre-Val de Loire
  - Hopital Nord Franche Comte, Belfort
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CH de DAX, Dax
  - CHU de DIJON, Dijon
  - CH Chartres, Le Coudray
  - Ch Du Mans, Le Mans
  - CHI Mont de Marsan, Mont-de-Marsan
  - CH de Saint-Lô, Saint-Lô
  - Hopital Foch, Suresnes
  - CHRU de TOURS, Tours